CLINICAL TRIAL: NCT04980469
Title: A Randomized, Double-blind, Placebo Controlled, Parallel Group Study to Explore the Effect of Vitex Negundo and Zingiber Officinale on Non-specific Chronic Low Back Pain Due to Sedentary Lifestyle
Brief Title: A Study to Explore the Effect of Vitex Negundo and Zingiber Officinale on Non-specific Chronic Low Back Pain Due to Sedentary Lifestyle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: EB/210402/VT/LBP
Record Dates: First submitted 2021-07-14; First posted 2021-07-28 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — ginger extract

STUDY DESIGN:
Intervention Model Description: Randomized, Double-blind, Placebo controlled, Parallel group
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitex negundo + Zingiber officinale (Experimental): Dosage: 200 mg/ Capsule;1 capsule twice daily Route: Oral
  Interventions: Other: Vitex negundo + Zingiber officinale
- Placebo (MCC) (Placebo Comparator): Dosage: 200 mg/ Capsule; 1 capsule twice daily Route: Oral
  Interventions: Other: Placebo (MCC)

INTERVENTIONS:
Other: Vitex negundo + Zingiber officinale — 200 mg/ Capsule
  Arms: Vitex negundo + Zingiber officinale
Other: Placebo (MCC) — 200 mg/ Capsule
  Arms: Placebo (MCC)

SUMMARY:
Clinical trial will study the effect of a formulation containing Vitex negundo leaf extract and Zingiber officinale extract on alleviating chronic low back pain and related disability in individuals leading a sedentary lifestyle. It will also evaluate the efficacy of the product on other factors associated with LBP, including mobility, work productivity and sleep quality.

DETAILED DESCRIPTION:
Vitex negundo is a large aromatic shrub or tree part of the family Lamiaceae. Many parts of the plant have been studied for their medicinal properties, as they contain phytochemicals and secondary metabolites in the plant leaves, roots, flowers, and seeds.

These bioactive compounds are the reason behind the plant's anti-inflammatory, antihistamine, anti-diabetic, anti-oxidant, anti-cancer and antimicrobial activity. In a study wherein the plant leaf extract was fed to rats, it revealed the pain relieving properties of the fresh Vitex negundo leaves, which could be mediated by prostaglandin synthesis inhibition. However, there are no clinical trials that use the plant for chronic low back pain relief. On the other hand, Zingiber officinale (ginger) is a part of the family Zingiberacae and is one of the most important medicinal plants in use today. It has been used for pain relief in both oral and topical forms. It has been used in clinical trials to alleviate pain during dysmenorrhea, muscle soreness, osteoarthritis and chronic low back pain. However, in the clinical trial studying its effect on chronic low back pain, ginger was used in the form of an aromatic oil.The use of both these extracts in all the studies mentioned saw minimal problems related to toxicity and are seen as safe for consumption without any harmful effects, especially due to their use in traditional medicine. It has been stated however that extremely high dosage of ginger could lead to gastrointestinal discomfort, central nervous system depression, allergic reactions, prolonged pre-existing bleeding, and arrhythmia.Therefore, this clinical trial will study the effect of a formulation containing Vitex negundo leaf extract and Zingiber officinale extract on alleviating chronic low back pain and related disability in individuals leading a sedentary lifestyle. It will also evaluate the efficacy of the product on other factors associated with LBP, including mobility, work productivity and sleep quality.

The present study is a randomized, double-blind, placebo controlled, parallel group study to explore the effect of Vitex negundo and Zingiber officinale on non-specific chronic low back pain due to sedentary lifestyle. Approximately 90 participants aged between ≥ 18 and ≤ 60 years will be screened. Both the IP and placebo trial arms will have atleast 30 completed participants after accounting for the screening failure and dropout/withdrawal rate of 20% each. The treatment duration for all the study participants will be 30 days.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged between 18 and 60 years old
2. Participants with a history of sub-acute low back pain with symptoms continuously persisting since ≥ 7 and ≤ 12 weeks.
3. Participants with pain of moderate to severe intensity (≥ 60 mm in the VAS) in the area between the 12 th ribs and the buttock creases.
4. Participants who have a Roland-Morris disability score between ≥ 8 and ≤ 15.
5. Participants with a Body mass index ≥ 20 and ≤ 35 kg/m 2 .
6. Participants with FBG ≤ 110 mg/ dl
7. Participants with TSH ≥0.40 and ≤ 4.2 mIU/L
8. Individuals physically inactive for ≥1/3 rd of wake time (barring only night sleep time), as determined using the Longitudinal Aging Study Amsterdam (LASA) sedentary behaviour questionnaire.
9. Participants who have given their signed Informed Consent.

Exclusion Criteria:

1. Participants currently undergoing treatment with analgesics of chemical (NSAIDS), animal or herbal origins
2. Participants currently undergoing treatment with any other muscle relaxant or any drugs having muscle relaxant properties
3. Participants with history suggesting off and on symptoms of low back pain since more than 12 months.
4. Individuals with history of structured physical exercise for ≥2 days/ week (includes but not limited to walking, jogging running, yoga or any other form of exercise).
5. Individuals with history of hyperacidity with atleast one episode/ week.
6. Participants with evidence of a clinically unstable disease, as determined by medical history, physical examination, that, in the Investigator's/medical monitor's opinion, preclude entry into the study.
7. Women who have undergone menopause i.e. Post- menopausal women
8. Participants with uncontrolled hypertension defined as systolic blood pressure ≥ 129 and/or diastolic blood pressure ≥ 89 mm Hg
9. Individuals with diagnosed cases of migraine
10. Participants who had spinal surgery within 1 year of study entry
11. Participants who have used steroids within 3 months of study entry or any other long-term treatment with steroids
12. Individuals with history of hypnotics use or other CNS depressants.
13. Participants with history of lumbar spinal stenosis, fibromyalgia, or ankylosing spondylitis
14. Participants who have severe scoliosis
15. Participants with more severe pain in a region other than the lower back
16. Participants with acute low back pain associated with chills or fever
17. Participants who are pregnant/breast feeding or are planning to get pregnant during the course of the study.
18. Individuals who have receives treatment with another investigational agent within the last 30 days.
19. Participants with known or suspected history of alcohol ordrug abuse based on medical history, physical examination, or the Investigators clinical judgment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2021-09-25 (Actual); Primary Completion 2022-02-07 (Actual); Study Completion 2022-02-07 (Actual)

PRIMARY OUTCOMES:
Roland Morris Questionnaire | Days 0, Day 7 and Day 30.
  To determine effect of 30 days administration of IP on functional activities due to low back pain as assessed by the change in Roland-Morris disability score from baseline as compared to the change in placebo. The scale is used to differentiate between patients who have chronic low back pain without any form of disability and those who experience some form of disability due to the pain experienced. Only participants with a Roland Morris disability score between ≥ 8 and ≤ 15 will be included in the study, to exclude individuals with minimal and extremely debilitating chronic low back pain.

SECONDARY OUTCOMES:
Fingertip-to-Floor Test | Days 0,and 30.
  Using this test, the forward bending flexibility and mobility of individuals with chronic low back pain will be assessed, as well as the impact of IP consumption on the same in comparison to placebo. Participants will be asked to bend forward and attempt to touch the floor with their fingertips. The investigator will then measure the distance between the floor and the participant's right long finger using a standard measuring tape. The difference in height between the floor and the participant's right long finger will be compared from baseline to Day 30, and in comparison to the placebo
Pain Visual Analogue Scale | Days 0, 7 and 30.
  Participants will be asked to recall the pain they experienced in the specified lower back region, after which they will be asked to mark a point on the 100-point visual analogue scale that corresponds to the level of pain experienced. Participants will have to self-administer the scale.
  minimum score 0 is referred to no pain at all and Maximum Score 100 is referred to as the worst possible pain
Work Productivity and Activity Impairment Questionnaire | Days 0,and 30.
  Chronic low back pain has been associated with lower work productivity in several studies. Using the Work Productivity and Activity Impairment Questionnaire, the impact of chronic low back pain on work and the performance of regular activities will be studied. The questionnaire consists of six questions, all the replies being categorized into 4 groups: 1) Percentage worktime missed, 2) Percentage impairment while working, 3) Percentage overall work impairment and 4) Percentage activity impairment.
Insomnia severity index | Days 0,and 30.
  Participants will be asked to recall their sleep patterns for the past month and then fill the aforementioned questionnaire on baseline and Day 30. In this study, the Change of insomnia severity due to chronic low back pain will be studied throughout the study duration from baseline and in comparison to placebo.
  The score ranges for the same are as follows:
  0-7: No clinically significant insomnia 8-14: Subthreshold insomnia 15-21: Clinical insomnia (moderate severity) 22-28: Clinical insomnia (severe)

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - Dr. Adkar clinic, Mumbai, Maharashtra
  - Shree Polyclinic, Mumbai, Maharashtra